CLINICAL TRIAL: NCT04187781
Title: Quality Control of CE-Certified Phonak Hearing Aids - 2019_34
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Sonova2019_34
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- external microphone old (Other)
  Interventions: Device: external microphone
- external microphone new (Other)
  Interventions: Device: external microphone

INTERVENTIONS:
Device: external microphone — External microphone is developed for direct transmission of speech into the hearing aids for better speech intelligibility, especially in noise.

SUMMARY:
Phonak Hearing Devices pass through different development and study phases. At an early stage, feasibility studies are conducted to investigate new algorithms, features and functions in an isolated manner. If the benefit is proven, their performance is then investigated regarding interdependency between all available algorithms, features and functions running in parallel in a hearing aid (pivotal/pre-validation studies) and, resulting from the pre-validation studies, they get optimized. Prior to product launch, the Phonak Hearing Systems get reviewed by a final quality control in terms of clinical trials. This is a validation study, investigating improved algorithms, features, functions and wearing comfort. This will be a clinical investigation which will be conducted mono centric at Sonova AG Headquarters based in Stäfa (Switzerland).

DETAILED DESCRIPTION:
This study will compare two settings of an external microphone under real life conditions with experienced hearing aid users.

The external microphone streams the signal (e.g. speaker) directly into the hearing instrument (HI).

The subject should rate the devices in the lab and after a hometrial. The comfort, regarding to the loudness and the sound quality will be tested with the two settings at home and in the lab. Also the speech intelligibility will be tested in the lab.

This will be a clinical investigation which will be conducted mono centric at Sonova AG Headquarters based in Stäfa (Switzerland).

ELIGIBILITY:
Inclusion Criteria:

* experienced hearing aid user
* severe hearing loss
* willingness and interest in testing an external microphone healthy outer ear
* willingness to wear behind the ear hearing aids
* Informed Consent as documented by signature

Exclusion Criteria:

* the audiogram is not in the fitting range of the intended hearing aid
* limited mobility and not in the position to attend weekly appointments in Stäfa (Switzerland)
* participant is not able to describe experiences and hearing impressions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
Rating of the subjective comfort for the old and the new setting | 6 weeks
  Rating of the comfort, regarding to the loudness, with the old and the new setting of the external microphone (%)

SECONDARY OUTCOMES:
Evaluation of the speech intelligibility in noise | 2 weeks
  Another Outcome measure of this study is the Evaluation of speech understanding in noise of the device with the old setting and the new setting. Speech understanding in noise will be evaluated with an objective and validated test procedure, the Outcome measure will be the speech intelligibility in %.
Subjective Sound Quality rating | 6 weeks
  The secondary Outcome measure of this study is the Evaluation of the perceived Sound Quality (rated via subjective satisfaction rating) of the signal with the old setting, compared to the new setting of the external microphone.
Subjective rating of natural sounds | 6 weeks
  The subject should rate in the hometrial how natural environmental sounds are with the hearing aids.

CONTACTS AND LOCATIONS:
Locations (1):
- Sonova AG, Stäfa, Switzerland